CLINICAL TRIAL: NCT06838390
Title: Microcurrent Versus Transcutaneous Electrical Nerve Stimulation on Pressure Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hajar Jamal Amin Mohammed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hajar-005204
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Pressure Area
Keywords: Micro current versus TENs on pressure ulcer
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Microcurrent therapy (Experimental): This group included 22 patients with pressure ulcer who received microcurrent therapy 8 weeks (3times /daily) in addition to their physical therapy program (circulatory exercise,stretching exercise, and ROM ex.) and medical treatment
  Interventions: Device: Microcurrent Therapy; Other: physical therapy program; Drug: medial treatment
- transcutaneous electrical nerve stimulation (Active Comparator): This group included 22 patients with pressure ulcers who received transcutaneous electrical nerve stimulation 8 weeks (3 times daily) in addition to their physical therapy program (circulatory exercise, stretching exercise, and range of motion exercise) and medical treatment.
  Interventions: Device: Transcutaneous electrical nerve stimulation; Other: physical therapy program; Drug: medial treatment

INTERVENTIONS:
Device: Microcurrent Therapy — The study uses a four-channel microcurrent therapy device to treat pressure ulcers. The treatment involves applying four electrodes to the area around the ulcer, ensuring microcurrent passage throughout the wound bed. The treatment is done three times a day, lasting 35-40 minutes. The microcurrents are delivered in a monophasic, pulsed, square-form wave pulse with a voltage of 21 mV, an intensity of 42 µA, and a current density of 4.2 µA/cm.
  Arms: Microcurrent therapy
Device: Transcutaneous electrical nerve stimulation — The study aimed to treat ulcers with TENS using a two-channel device, delivered three times a day, for 8 weeks. The device induced peripheral vasodilation and activate local blood flow, potentially promoting wound healing. The treatment was delivered using a pulse train duration of 300 ms, with an internal frequency of 100 Hz and a burst frequency of 2 Hz.
  Arms: transcutaneous electrical nerve stimulation
Other: physical therapy program — The physiotherapy program included circulatory circulatory exercises, stretching exercises, and ROM exercises.
Drug: medial treatment — patients was given their drugs from their physicians

SUMMARY:
The purpose of the study was to evaluate which is more effective, microcurrent or transcutaneous electrical nerve stimulation, in treating pressure ulcers in elderly patients.

DETAILED DESCRIPTION:
* Pressure sores are common problems in today's health care. A pressure sore leads to physiological as well as psychological suffering for the individual affected. The cost for the society, associated with prevention and treatment of pressure sores, is considerable
* Furthermore, the need for this study was developed from the lack of quantitative knowledge and information in the published studies about the effect of microcurrent and transcutaneous electrical nerve stimulation in treating pressure ulcers in elderly patients.
* This study will be carried out to provide guidelines about the effectiveness of microcurrent and transcutaneous electrical nerve stimulation in treating pressure ulcer and to assist in planning an ideal treatment regimen to increase healing of pressure ulcers in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

Subject selection was done according to the following criteria:

* Age range between 40 and 60 years.
* Male and female patients will participate in the study.
* All patients enrolled in the study had their informed consent.
* Pressure ulcer grades were grade II and III.
* A relative or legal tutor provided consent when participants were incapable of making decisions.
* The trial complied with the ethical principles of the Helsinki Declaration for medical research in humans.
* Pressure ulcers were located in the sacral area

Exclusion Criteria:

* Age less than 40 years or more than 60 years
* A cardiac pacemaker or another implanted electric device.
* Cognitive problems or hearing loss.
* Pre-existing joint disorder before pressure ulcer.
* Patients who have co-morbidities such as diabetes mellitus, rheumatoid arthritis, hypertension, and cardiac and renal patients,
* Osteosynthesis implants near the ulcer, pressure ulcers in the occipital region, cancer, and osteomyelitis.
* Abnormal blood markers at baseline indicating limited healing potential (anemia, iron deficit, protein deficit, dehydration, non-controlled diabetes, or hypothyroidism).
* Allergy to the usual treatment for ulcer healing, systemic infection, and ulcer treatment with growth factor or vacuum-assisted closure in the 30 days before the Trial

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Assessment of ulcers length x width using Pressure Ulcer Scale for Healing | at baseline and after 8 weeks
  The Pressure Ulcer Scale for Healing is a tool used to measure ulcer healing. It assesses the length x width of the ulcer (measuring the greatest length-head to toe-and the greatest width-side to side-using a centimeter ruler). It scores from 0-surface area of 0 cm²-to 10-surface area >24 cm²); The total score of pressure ulcer healing is calculated by adding three sub-scores, ranging from 0 (completely healed) to 17 (worst wound state), and comparing it at each time point indicates improvement or deterioration.
Assessment of ulcers exudate amount using Pressure Ulcer Scale for Healing | at baseline and after 8 weeks
  The Pressure Ulcer Scale for Healing is a tool used to measure ulcer healing.It assesses exudate amount (classified as none: score 0; light: score 1; moderate: score 2; or heavy: score 3); The total score of pressure ulcer healing is calculated by adding three sub-scores, ranging from 0 (completely healed) to 17 (worst wound state), and comparing it at each time point indicates improvement or deterioration.
Assessment of ulcers tissue type using Pressure Ulcer Scale for Healing | at baseline and after 8 weeks
  The Pressure Ulcer Scale for Healing is a tool used to measure ulcer healing. It assesses tissue type (score 1: superficial wound with epithelial tissue; score 2: the wound is clean and contains granulation tissue; score 3: there is any amount of slough present; score 4:necrotic tissue is present). If the wound is closed, the score is 0.
  The total score of pressure ulcer healing is calculated by adding three sub-scores, ranging from 0 (completely healed) to 17 (worst wound state), and comparing it at each time point indicates improvement or deterioration.

SECONDARY OUTCOMES:
Evaluation of blood flow in both the major and the minor vessels of the body. | at baseline and after 8 weeks
  Medical Doppler ultrasound is used in clinical adjustments to evaluate blood flow in major and minor vessels. It shows normal and abnormal sign waveforms using spectral Doppler technique, which is individual to each vessel. Understanding normal and abnormal diagnostics is crucial for operators and clinicians

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No